CLINICAL TRIAL: NCT00105118
Title: 10 Hz rTMS to Subject Specific Regions of Cerebral Cortex Improves Memory in Healthy Subjects
Brief Title: Effect of Transcranial Magnetic Stimulation on Memory
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050100; 05-M-0100
Record Dates: First submitted 2005-03-04; First posted 2005-03-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-02

CONDITIONS: Healthy; Healthy Volunteer; HV
Keywords: Cognition; Alpha; Schizophrenia; Functional Connectivity; Oscillatory Potential
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Device: Magstim Super Rapid Magnetic Stimulator

SUMMARY:
This study will examine the effect of transcranial magnetic stimulation (TMS) on short-term memory in healthy adults. Healthy people use their brains to answer short-term memory questions in a different way than do patients with schizophrenia. Attention and memory deficits in schizophrenia patients significantly hamper their recovery and rehabilitation, yet there are no effective treatments for these impairments. TMS is a method of brain stimulation that may be able to change the electrical activity of the nerve cells of the brain and improve certain brain functions. This study will explore the effect of TMS on memory and perhaps discover brain processes that may be helpful in developing new ways to treat schizophrenia.

Healthy volunteers between 18 and 55 years of age, excluding pregnant women, may be eligible for this study. Participants undergo the following tests and procedures:

* Medical history, physical examination, blood tests, electrocardiogram (EKG), and urine pregnancy test for women of childbearing age.
* Magnetic resonance imaging (MRI) and functional MRI (fMRI). These tests are done in participants who have not had structural and functional MRIs as participants in NIMH's 2-day schizophrenia study within 90 days of entering the current study. MRI is done to locate the place in the brain to simulate with TMS and fMRI is done to look at brain activity while the subject solves short-term memory tasks. Both tests are done at the same session. Before the scan, four vitamin E capsules are taped to the subject's scalp. After the capsules are in place, the subject lies on a stretcher that is moved into the scanner - a narrow cylinder with a strong magnetic field. During the scan, subjects are asked to do some simple tests, such as watching pictures on a screen or pressing buttons in response to numbers they were shown a few seconds earlier. Scanning may take up to 2 hours, but usually lasts between 45 and 90 minutes.
* TMS. For this procedure, subjects receive either active TMS or a sham procedure (placebo) that imitates TMS but does not use real electrical stimulation. For TMS, an insulated wire coil is placed on the scalp and a brief electrical current is passed through it. This generates magnetic pulses that travel through the scalp and skull and cause small electrical currents in the cortex, or outer part of the brain. The stimulation may cause muscle twitching in the scalp or face and may also cause small movement of the limbs. During the procedure, electrodes are taped to the scalp to record the electrical activity of the brain while short-term memory is tested. Two tests make up a set. There are a total of six test sets; each set takes about 3 minutes. Five periods of electrical stimulation are delivered before each test set. Each period of stimulation lasts 5 seconds, followed by a 10-second rest period. The stimulation-rest intervals continue until five periods of TMS have been applied. For the memory test, subjects press a key on a computer keyboard as quickly and accurately as possible in a test of their ability to remember a string of numbers, or letters.
* Questionnaires. At the beginning and end of the TMS session, participants fill out questionnaires that assess their mood, ability to concentrate, and level of anxiety.

DETAILED DESCRIPTION:
Psychiatrists have recognized cognitive dysfunction as the principal impediment to recovery and psychosocial rehabilitation of patients with schizophrenia since the first edition of Emil Kraepelin's 1893 masterwork, Dementia Praecox. While currently available pharmacotherapy may improve psychotic symptoms, there is still no largely effective treatment for impairments of critical executive functions - attention and working memory - that are widely considered the functional nexus of this extremely costly illness. Thus, it appears heuristically reasonable to consider putative modes of treatment that may specifically target these deficits. For example, abundant evidence supports the assumption that pre-task alpha band power, measured as mean peak frequency, is inversely associated with reaction time (RT) - an index of encoding efficiency - in a working memory task. Additionally, recent evidence suggests pre-task alpha peak frequency predicts outcome on tests of working memory. Evidence also suggests patient with schizophrenia have low pre-task alpha peak frequency, and slower RT on working memory paradigms, such as the n-back and Sternberg compared with healthy controls; taken together, the weight of evidence lends plausibility to the assumption that an increase in patients' pre-task alpha band power might be associated with a faster reaction time. Notably in this regard, recent evidence suggests transcranial magnetic stimulation (TMS) may increase pre-task alpha, and is associated with a faster RT in healthy subjects. There are as yet no reports of the effect of TMS on alpha band peak frequency, or reaction time, in patients with schizophrenia. A critical obstacle to progress in the clinical neuroscience of TMS effects in human subjects until now has been the absence of a means to determine the optimal subject-specific brain region to target with TMS. Cortical targets for stimulation are customarily selected on the basis of group mean data, with the tacit assumption that candidates for TMS all utilize the same distributed neural circuit to perform a particular cognitive task. This untested assumption is a conceivable source of the confusing discrepancy of TMS clinical trial outcomes, for example, in the depression treatment literature. In this regard, a group from our laboratory recently reported the use of structural equation modeling (SEM) based path analysis to construct group and subject-specific models of the 2-back working memory task in healthy subjects studied with PET. The results of this investigation suggest there may be a significant association between cognitive strategy, circuit path, and memory performance. We found higher scores were associated with activation of a left hemisphere distributed circuit, and a verbal cognitive strategy, while lower scoring subjects utilized a right hemisphere circuit, and a visuo-spatial strategy. Notably, these findings are congruent with those of previous studies that used different methods of analysis and a similar paradigm. Taken together, these data suggest that a trial of TMS aimed at improving working memory reaction time by elevating pre-task alpha power should first identify the predominant nodes of a subject-specific working memory sub-network as putative sites of stimulation. There are no reports of such an approach to TMS target selection in either healthy controls, or patients with schizophrenia. In this proof of concept with healthy subjects protocol, our principle assumption is alpha frequency TMS directed to a subject-specific predominant node (right or left DLPFC) of a distributed neural network reduces reaction time on the n-back and Sternberg working memory paradigms.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male and Female subjects, age 18-55

EXCLUSION CRITERIA:

1. Significant psychiatric, or severe chronic medical illness at the time of the study, or by history. This criterion includes the absence of substance abuse histories, learning disabilities or any other DSM-IV AXIS I or II disorder with documented cognitive impairment. The P.I. or his designate will evaluate medical histories. Medical conditions that are judged not to interfere with the study may be allowed.
2. Pregnancy, personal or family history of epilepsy, concurrent use of tricyclic antidepressants, neuroleptic agents, or any licit or illicit drugs that could lower the seizure threshold, or history of complicated migraine.
3. Persons with surgically or traumatically implanted ferro-magnetic objects in the head that may pose a physical hazard during magnetic stimulation will also be excluded.
4. Use of psychotropic substances in the last 3 months.
5. Head injury with a period of more than 15 minutes unconsciousness, or head trauma with any duration loss of consciousness in the last year, or any evidence of functional impairment due to and persisting after head trauma.
6. Use of caffeine or tobacco in the 2 hours preceding the test.
7. Subjects who have been previously excluded from NIH MRI or TMS protocols for safety reasons.
8. Subjects who are found to have eye lesions on exam.
9. First degree relative with a history of cognitive disorder with onset before age 55 by subject report, and by collateral report of at least one other family member, if necessary.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2005-03; Study Completion 2006-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] McGurk SR, Mueser KT. Cognitive functioning and employment in severe mental illness. J Nerv Ment Dis. 2003 Dec;191(12):789-98. doi: 10.1097/01.nmd.0000100921.31489.5a. PMID 14671455
- [Background] McGurk SR, Moriarty PJ, Harvey PD, Parrella M, White L, Davis KL. The longitudinal relationship of clinical symptoms, cognitive functioning, and adaptive life in geriatric schizophrenia. Schizophr Res. 2000 Mar 16;42(1):47-55. doi: 10.1016/s0920-9964(99)00097-3. PMID 10706985
- [Background] Docherty NM, Hawkins KA, Hoffman RE, Quinlan DM, Rakfeldt J, Sledge WH. Working memory, attention, and communication disturbances in schizophrenia. J Abnorm Psychol. 1996 May;105(2):212-9. doi: 10.1037//0021-843x.105.2.212. PMID 8723002